CLINICAL TRIAL: NCT04941690
Title: Prevalence and Correlates of Erectile Dysfunction, Psychological Disorders, and Sexual Performance Among Men Seeking Medical Help for Preconception Test, Infertility and Wife Miscarriage
Brief Title: Erectile Dysfunction, Psychological Disorders, and Sexual Performance Among Men Seeking Medical Help for Fertility
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Yu xiaowei, Clinical Professor, Center for Reproductive Medicine and Center for Prenatal Diagnosis, The First Hospital of Jilin University
Other Study IDs: 21K064-001
Record Dates: First submitted 2021-06-21; First posted 2021-06-28 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Erectile Dysfunction; Sexual Dysfunction; Premature Ejaculation; Infertile Men; Fertile Men; Wife's Miscarriage
MeSH Terms: conditions — Erectile Dysfunction; Sexual Dysfunction, Physiological; Premature Ejaculation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Men seen for preconception physicals: Ready to conceive, i.e. not having contraception and not having children for less than 1 year
  Interventions: Other: A questionnaire method was used.
- Men seen for infertility: Couples who have not used contraception and have not had children for more than 1 year
  Interventions: Other: A questionnaire method was used.
- Men who visited the clinic for their wives' miscarriage: Couples whose wives were previously pregnant but terminated the pregnancy due to fetal abortion, spontaneous abortion, biochemical pregnancy, fetal malformation or ectopic pregnancy
  Interventions: Other: A questionnaire method was used.

INTERVENTIONS:
Other: A questionnaire method was used. — The questionnaire included general population information, International Index of Sexual Function-5 (IIEF-5), Premature Ejaculation Diagnostic Tool (PEDT), General Anxiety Disorder-7 and CPSI.

SUMMARY:
According to the World Health Organization (WHO) and the World Association for Sexual Health (WAS), sexual health is directly related to everyone's mental health and quality of life. Sexuality is innate to humans and is closely linked to their reproduction. Thus, a correlation between unmet fertility desires and sexual disorders can be observed in infertile couples. In fact, sexual intercourse itself will not be as natural in most cases and will preferentially occur during the "reproductive window". Thus, sexuality will be deprived of recreational and erotic activities, and sexuality will be used only for reproduction. For many men, sexual intercourse will become coercive, repetitive and mechanical, offering little emotion.

The interactions between infertility and wife recurrent miscarriage in sexuality are numerous and complex. Many men will perceive their infertility as a loss of masculinity and virility and may feel low self-esteem and depression, in addition, Decreased sperm quality may lead to anxiety in men, which may eventually lead to temporary Sexual Dysfunction (SD).Therefore, the need to identify SD and its severity is crucial for infertile men before receiving individualized male treatment.

DETAILED DESCRIPTION:
In this study, a cross-sectional and clinical survey was conducted using a questionnaire method in the male department of the reproductive center of the First Hospital of Jilin University, China. The questionnaire included general population information, International Index of Sexual Function-5 (IIEF-5), Premature Ejaculation Diagnostic Tool (PEDT), General Anxiety Disorder-7 and CPSI. The inclusion criteria were: 1, men living with their wives and planning to have children; 2, men seeking medical help for preconception tests, infertility, and recurrent miscarriage of their wives; and 3, consenting to participate in the survey and signing an informed consent form. Exclusion criteria were: 1, men with significant genital malformations, severe cardiovascular disease, stroke and mental disorders; 2, men who could not live with their female partners every day because they worked in different cities; 3, medical history of female partners with reproductive system abnormalities by gynecological examination.

Investigators also collect relevant test results (if any) from the included patients during the visit. All patients routinely undergo a detailed male examination; for patients with preconception testing, the examination may include sperm quality, blood group, infection items (hepatitis B, hepatitis C, syphilis, AIDS), TORCH, etc; For infertile patients, only a sperm quality is performed in the first step; For patients whose wives have had recurrent miscarriages and are preparing to conceive again, the examination may include a detailed male examination, sperm quality, Chromosomes, blood group, infections (hepatitis B, C, syphilis, AIDS), TORCH, etc. If no abnormality is found, there is no follow-up examination, and if there is abnormality, further follow-up examination will be performed according to the process of Chinese Male Disease Diagnosis and Treatment Guidelines (2016). All consultations are in accordance with the process of Chinese Male Disease Diagnosis and Treatment Guidelines (2016). This study will not increase the physical and financial burden of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* 1, men living with their wives and planning to have children; 2, men seeking medical help for preconception tests, infertility, and recurrent miscarriage of their wives; and 3, consenting to participate in the survey and signing an informed consent form.

Exclusion Criteria:

* 1, men with significant genital malformations, severe cardiovascular disease, stroke and mental disorders; 2, men who could not live with their female partners every day because they worked in different cities; 3, medical history of female partners with reproductive system abnormalities by gynecological examination.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: men seeking medical help for preconception tests, infertility, and recurrent miscarriage of their wives
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-06-26 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Occurrence of sexual dysfunction among men seen for preconception testing, infertility, and wife miscarriage | 12-26-2021
  Evaluation of the occurrence of sexual dysfunction among men seen for preconception testing, infertility, and wife miscarriage, A questionnaire method was used.
  The questionnaire included general population information, International Index of Sexual Function-5 (IIEF-5), Premature Ejaculation Diagnostic Tool (PEDT), General Anxiety Disorder-7 and CPSI.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Reproductive Medicine and Center for Prenatal Diagnosis, Jilin University First Hospital, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided